CLINICAL TRIAL: NCT03632590
Title: The Effects of Magnesium Salts on Vascular Stiffness: A Randomized Controlled Trial in Healthy Overweight and Slightly Obese Men and Women
Brief Title: Magnesium and Vascular Stiffness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Nedmag Industries Mining and Manufacturing B.V. (Unknown)
Responsible Party: Principal Investigator, Stephan J.L. Bakker, Prof. dr., University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: METc2017/220
Record Dates: First submitted 2018-08-06; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Vascular Stiffness; Blood Pressure
Keywords: Magnesium; Supplements
MeSH Terms: interventions — magnesium citrate; Magnesium Sulfate; Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Magnesium Citrate (Experimental): 450 mg of Magnesium Citrate per day
  Interventions: Dietary Supplement: Magnesium Citrate
- Magnesium Sulfate (Experimental): 450 mg of Magnesium Sulfate per day
  Interventions: Dietary Supplement: Magnesium Sulfate
- Magnesium Oxide (Experimental): 450 mg of Magnesium Oxide per day
  Interventions: Dietary Supplement: Magnesium Oxide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium Citrate — 450 mg of Magnesium Citrate per day (6 capsules per day) for 24 weeks
  Arms: Magnesium Citrate
Dietary Supplement: Magnesium Sulfate — 450 mg of Magnesium Sulfate per day (6 capsules per day) for 24 weeks
  Arms: Magnesium Sulfate
Dietary Supplement: Magnesium Oxide — 450 mg of Magnesium Oxide per day (6 capsules per day) for 24 weeks
  Arms: Magnesium Oxide
Drug: Placebo — The placebo capsules will contain starch (Amylum solani) for 24 weeks
  Arms: Placebo

SUMMARY:
This four-arm randomized controlled trial was designed to study the effects of magnesium supplements (total daily dose: 450 mg elemental magnesium) on vascular stiffness in healthy overweight and slightly obese men and women. In addition, the effects of magnesium supplements on blood pressure and gut microbiota will be evaluated. Three groups will receive magnesium supplements (magnesium oxide, magnesium citrate or magnesium sulphate) and one group will receive a placebo.

DETAILED DESCRIPTION:
Observational epidemiologic studies have observed an inverse relationship between daily dietary magnesium intake and blood pressure. Except for blood pressure, magnesium may also beneficially affect other cardiovascular risk markers. Whether all these effects translate into improved vascular function is not known. Different vascular function markers at various stages on the pathway between diet and disease exist. One of these markers, vascular stiffness, is closely related to the process of atherosclerosis, an independent cardiovascular risk factor, and predictive of future cardiovascular events and mortality. A recently published intervention study showed that oral magnesium citrate supplementation of 350 mg per day for 24 weeks was well-tolerated and improved vascular stiffness by 1.0 m/s. Importantly, it was not established whether the beneficial effect on vascular stiffness was due to the supplementation of magnesium or due to citrate. This may involve effects on gut microbiota and systemic metabolic effects. The current study was designed to (1) reproduce the result of the earlier study and to (2) investigate whether there is a difference between different commonly used magnesium salts (magnesium citrate, magnesium sulphate and magnesium oxide) in terms of effects on vascular stiffness, blood pressure and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 45-70 years
* Women postmenopausal: two or more years after last menstruation
* BMI between 25-35 kg/m2 (overweight and slightly obese)
* Plasma glucose < 7.0 mmol/L
* Serum total cholesterol < 8.0 mmol/L (further testing is recommended for excessive hyperlipidemia (serum total cholesterol ≥ 8.0 mmol/L) according to the Standard for cardiovascular risk management of the Dutch general practitioners community (NHG))
* Serum triacylglycerol < 4.5 mmol/L (Friedewald formula)
* No current smoker
* No diabetic patients
* No familial hypercholesterolemia
* No abuse of drugs
* Less than 21 alcoholic consumptions per week
* Stable body weight (weight gain or loss <3 kg in the past three months)
* No use of proton pump inhibitors
* No use of magnesium supplements
* No severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* No active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebro vascular accident
* Willingness to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study and during the study
* No difficult venipuncture as evidenced during the screening visit
* Written informed consent

Exclusion Criteria:

* High habitual dietary magnesium intake (defined as urinary magnesium excretion of 7.0 or 5.9 mmol/24-h or more for men and women, respectively)
* Plasma glucose ≥ 7.0 mmol/L
* Serum total cholesterol ≥ 8.0 mmol/L
* Serum triacylglycerol ≥ 4.5 mmol/L
* Current smoker, or smoking cessation <12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 21 alcoholic consumptions per week
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Use of proton pump inhibitors
* Use of magnesium supplements
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebro vascular accident
* Not willing to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study and during the study
* Not or difficult to venipuncture as evidenced during the screening visit

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in vascular stiffness | Baseline, FU-1 (2 weeks), FU-2 (12 weeks), and FU-3 (24 weeks)
  Measured from carotid-femoral pulse wave velocity (PWV). For this assessment, a SphygmoCor will be used (SphygmoCor v9, AtCor Medical).

SECONDARY OUTCOMES:
Change in blood pressure | Baseline, FU-1 (2 weeks), FU-2 (12 weeks), and FU-3 (24 weeks)
  Measured from a semi continuous blood pressure monitoring device
Change in gut microbiota | Baseline, FU-1 (2 weeks), FU-2 (12 weeks), and FU-3 (24 weeks)
  Measured from fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Stephan JL Bakker, MD-PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Schutten JC, Joris PJ, Groendijk I, Eelderink C, Groothof D, van der Veen Y, Westerhuis R, Goorman F, Danel RM, de Borst MH, Bakker SJL. Effects of Magnesium Citrate, Magnesium Oxide, and Magnesium Sulfate Supplementation on Arterial Stiffness: A Randomized, Double-Blind, Placebo-Controlled Intervention Trial. J Am Heart Assoc. 2022 Mar 15;11(6):e021783. doi: 10.1161/JAHA.121.021783. Epub 2022 Mar 5. PMID 35253448
- [Derived] Schutten JC, Joris PJ, Mensink RP, Danel RM, Goorman F, Heiner-Fokkema MR, Weersma RK, Keyzer CA, de Borst MH, Bakker SJL. Effects of magnesium citrate, magnesium oxide and magnesium sulfate supplementation on arterial stiffness in healthy overweight individuals: a study protocol for a randomized controlled trial. Trials. 2019 May 28;20(1):295. doi: 10.1186/s13063-019-3414-4. PMID 31138315